CLINICAL TRIAL: NCT04125186
Title: Epidemiology and Burden of Nocturia Due to Nocturnal Polyuria in the United States: The EpiNP Study
Brief Title: A Cross-Functional, Population-Representative, Web-Based, Epidemiologic Study to Estimate the Prevalence and Burden of Nocturia Due to Nocturnal Polyuria in the US
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EVA-21176
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2020-08

CONDITIONS: Nocturnal Polyuria
Keywords: Bladder diary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pilot Part: After providing consent, participants with nocturia will complete web-based baseline EpiNP survey followed by 3-day bladder diary and then a qualitative interview.
  Interventions: Diagnostic Test: Testing of EpiNP baseline survey, bladder diary and a qualitative interview; Other: No other intervention
- Main Part: After providing consent, participants will complete web-based baseline EpiNP survey. All respondents who report greater than equal to (≥)2 voids/night, and a randomly selected cohort of respondents reporting 0 and 1 void/night will use the EpiNP 3-day web-based bladder diary.
  Interventions: Diagnostic Test: Baseline EpiNP survey; Diagnostic Test: Bladder diary; Other: No other intervention

INTERVENTIONS:
Diagnostic Test: Baseline EpiNP survey — The survey takes approximately 20 to 30 minutes to complete, and consists of the following: Short Form Health Survey version 2.0 (SF-12v2.0); Lower Urinary Tract Symptoms (LUTS) Tool; Patient Perception of Bladder Condition (PPBC); Self-report Medical History and Current Medication Form; Nocturia Impact Diary (NID); Disease-Specific Healthcare-Seeking Behavior and Treatment; Epworth Sleepiness Questionnaire (ESS); Patient Reported Outcome Measurement Information System Fatigue-Short Form version 1.0 (PROMIS F-SFv1.0); Patient Health Questionnaire (PHQ-8); Work Productivity and Activity Index (WPAI-SHP); Sexual health questions; lifestyle and sociodemographic questions; additionally, only men will complete the International Prostate Symptom Score (IPSS).
  Groups: Main Part
Diagnostic Test: Bladder diary — It consists of four components: measurement of waist and neck circumference, daily voiding diary (to assess voiding patterns, including frequency, volume, associated urgency, and incontinence episodes over a 24-hour period), NID (to assess nocturia impact), and assessment of morning sleepiness for 3 consecutive days and nights (including the morning of the fourth day).
  Groups: Main Part
Diagnostic Test: Testing of EpiNP baseline survey, bladder diary and a qualitative interview — This part briefly reviews the usability of the EpiNP survey and bladder diary. The feedback obtained after qualitative interview will be used to refine and finalize the instructions sent to the participants in the main part.
  Groups: Pilot Part
Other: No other intervention — No other intervention

SUMMARY:
To estimate the prevalence of nocturia due to nocturnal polyuria (NP) in the US and describe the demographic and clinical characteristics as well as the burden of illness in participants with nocturia due to NP.

ELIGIBILITY:
Inclusion Criteria:

* At least 30 years of age;
* Willing to provide informed consent;
* Able to read US-English or Spanish
* Able to use a computer and access the internet.

Exclusion Criteria:

* Symptomatic acute urinary tract infection (UTI) (experiencing symptoms such as pain or burning when you urinate, strong and frequent urge to urinate, or cloudy, bloody, or strong-smelling urine);
* Currently pregnant or ≤12 months postpartum;
* Recent surgery in the last <6 months;
* Current lifestyle that leads to irregular or atypical circadian patterns (e.g. employed in overnight shift work)
* Prior YouGov survey participation in past two weeks

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in two parts: (1) Pilot part: approximately 30 participants who have a physician diagnosis of nocturia. Participants will be recruited by one clinical site in the US. (2) Main part: a sample of 10,000 participants who are representative of the general population in the US stratified by age (≥30), gender, and race. Participants will be recruited by e-mail from a web-based panel of people that have previously opted in to be contacted for research studies.
Sampling Method: Probability Sample
Enrollment: 10190 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of nocturia due to NP, NP with overactive bladder (OAB), NP with benign prostatic hyperplasia (BPH), and NP with BPH/OAB | Between July 2019 and June 2020
  Nocturia due to NP will be derived using data of participants who completed the 3-day bladder diaries. Nocturnal polyuria was defined when nocturnal urine production proportional to daytime urine production was greater than threshold 0.33 (Nocturnal Polyuria index [NPi]). Prevalence will be calculated using number of participants with nocturia due to NP, in the numerator (overall and by relevant strata [e.g., by age/race/gender categories]), with publicly-available estimates of the US population in the denominator (overall and for relevant strata). In addition, the prevalence of NP with OAB, NP with BPH, and NP with BPH/OAB will also be estimated.
To describe and compare demographic and clinical characteristics in participants with nocturia due to NP, NP with OAB, NP with BPH, and NP with BPH/OAB | Between July 2019 and June 2020
To describe and compare burden of illness in participants with nocturia due to NP, NP with OAB, NP with BPH, and NP with BPH/OAB | Between July 2019 and June 2020
  The burden measures (including health-related quality of life [HRQL], work productivity, fatigue, sleep, and depression as assessed through EpiNP survey and bladder diary) in participants with nocturia due to NP, NP with OAB, NP with BPH, and NP with BPH/OAB (overall and by relevant strata [e.g., by age/race/gender categories]) will be presented.

SECONDARY OUTCOMES:
Prevalence of nocturia due to NP across the subgroups of respondents | Between July 2019 and June 2020
  Before using 3-day bladder diary in main part, the responders of the baseline EpiNP survey were stratified by three subgroups: all respondents who report ≥2 voids/night, randomly selected cohort of respondents reporting 0 and 1 void/night. Prevalence will be calculated using number of participants with nocturia due to NP across the subgroups of respondents, in the numerator, with publicly-available estimates of the US population in the denominator.
To describe and compare demographic and clinical characteristics in participants with nocturia due to NP across the subgroups of respondents | Between July 2019 and June 2020
To describe and compare burden of illness in participants with nocturia due to NP across the subgroups of respondents | Between July 2019 and June 2020
  Before using 3-day bladder diary in main part, the responders of the baseline EpiNP survey were stratified by three subgroups: all respondents who report ≥2 voids/night, randomly selected cohort of respondents reporting 0 and 1 void/night. The burden measures will be compared across the subgroups of respondents who self- report either 0 or 1 void/night with those reporting ≥2 voids/night.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Evidera Inc., Seattle, Washington, United States

REFERENCES:
- [Result] Weiss JP, Bosch JLHR, Chapple CR, Bacci ED, Simeone JC, Rosenberg MT, Mueller ER, Andersson FL, Juul K, Chughtai B, Coyne KS. The Prevalence of Nocturnal Polyuria in the United States: Results from the Epidemiology of Nocturnal Polyuria Study. Eur Urol Focus. 2022 Sep;8(5):1415-1423. doi: 10.1016/j.euf.2021.12.016. Epub 2022 Jan 14. PMID 35039242
- [Result] Bosch JLHR, Chapple CR, Mueller ER, Rosenberg MT, Chughtai B, Juul K, Coyne KS, Andersson FL, Bacci ED, Simeone JC, Weiss JP. Differences in the Prevalence of Nocturnal Polyuria in the U.S. by Definition: Results from the Epidemiology of Nocturnal Polyuria Study. J Urol. 2022 Jul;208(1):144-154. doi: 10.1097/JU.0000000000002500. Epub 2022 Apr 21. PMID 35446110
- [Result] Chapple CR, Rosenberg MT, Mueller ER, Chughtai B, Weiss JP, Juul K, Brooks AB, Bacci ED, Andersson FL, Coyne KS, Bosch JR. The patient burden of nocturnal polyuria in the United States: Results from the epidemiology of nocturnal polyuria (EpiNP) study. Neurourol Urodyn. 2023 Mar;42(3):573-585. doi: 10.1002/nau.25126. Epub 2023 Jan 19. PMID 36655731
- [Result] Mueller ER, Weiss JP, Bosch JLHR, Chughtai B, Rosenberg MT, Bacci ED, Simeone JC, Andersson FL, Juul K, Coyne KS, Chapple CR. Nocturnal polyuria in women: results from the EpiNP study. Int Urogynecol J. 2023 Aug;34(8):1743-1751. doi: 10.1007/s00192-022-05432-x. Epub 2023 Jan 28. PMID 36708403